CLINICAL TRIAL: NCT02767258
Title: Randomized Clinical Trial: Effect of Nursing Interventions on Prevention of Dry Eye in Critically Ill Patients
Brief Title: Effect of Nursing Care on Prevention of Dry Eye
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diego Dias de Araújo (Other)
Collaborators: State University of Montes Claros (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Diego Dias de Araújo, Teacher and Student Doctoral Nursing, Federal University of Minas Gerais
Organization: Federal University of Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EE/UFMG
Record Dates: First submitted 2016-05-06; First posted 2016-05-10 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye; Diseases of the eye and adnexa
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Comparator: Eye drop (Active Comparator): Eye drop LACRIBELL® - two drops each eye, two times a day, after eye cleansing.
  Interventions: Device: LACRIBELL®
- VIDISIC® GEL (Experimental): Ocular gel VIDISIC® GEL applied two times a day at the lower palpebra from medium line to the lateral border.
  Interventions: Device: VIDISIC® GEL

INTERVENTIONS:
Device: LACRIBELL® — Hypromellose and dextran based eyedrop, used in the treatment of dry eye.
  Other Names: liquid artificial tears; eyedrop
  Arms: Sham Comparator: Eye drop
Device: VIDISIC® GEL — Carbomer based gel, used in the treatment of dry eye.
  Other Names: artificial tear gel
  Arms: VIDISIC® GEL

SUMMARY:
Clinical trial for prevention, randomized controlled, parallel, double-blind, with three arms, which purpose is verify the nursing interventions (artificial tear gel and liquid artificial tears)effects to prevent dry eye in adult patients admitted in ICU.

DETAILED DESCRIPTION:
Critically ill patients are at higher risk for dry eye and the mechanisms responsible for ocular lubrication and protection can be compromised. However, the literature diverges on which is the best clinical practice for treatment. Thus, the general objective of this study was to evaluate the risk for developing dry eye in critically ill patients and the effectiveness of three types of interventions: eye gel and eyedrops (control group). The specific objectives were: verify the most effective intervention for the prevention of dry eye from the available literature and provided by: eye gel compared to the control group eyedrops who received eye care through randomized controlled clinical trial. Patients and methods: This study is a randomized controlled trial to determine the best care for the prevention of dry eye from those available on the market (eye drops and eye gel), in the period from 14/01/2016 to 31/12/2019 . The expected result is: negative values in Schirmer test and no corneal ulcers presence.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years;
* Did not present dry eye at the time of admission;
* Stay in the ICU for at least 24 hours;
* Be in mechanical ventilation therapy;
* Glance less than 5 per minute;
* Comatose, sedated or Glasgow less than or equal to 7;
* Consent to participate in research or have.

Exclusion Criteria:

* Have not the responsabille authorization;
* Patients with severe eye disease or with history of adverse effects after use of any of the interventions proposed and not tolerate the treatment: artificial tear gel, artificial tear liquid and saline 0.9%.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Dry Eye | Five consecutive days
  Interventions will be applied in both eyes of the patients from 12 to 12 hours for five consecutive days. Schirmer test will be applyed to evaluate the lacrimal volume. Fluorescein test will be applyed to evaluate the ocular surface.

CONTACTS AND LOCATIONS:
Overall Officials: Diego D Araújo, PhD student, Principal Investigator — State University of Montes Claros, Minas Gerais, Brazil
Locations (1):
- Santa de Misericórdia Montes Claros, Montes Claros, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
The study and the information provided will be confidential and used only for purposes of this research. Disclosure of information will be anonymous and in conjunction with the responses of a group of people, never individually.

REFERENCES:
- [Background] de Araujo DD, Almeida NG, Silva PM, Ribeiro NS, Werli-Alvarenga A, Chianca TC. Prediction of risk and incidence of dry eye in critical patients. Rev Lat Am Enfermagem. 2016;24:e2689. doi: 10.1590/1518-8345.0897.2689. Epub 2016 May 17. PMID 27192415